CLINICAL TRIAL: NCT02060682
Title: Post-Market Registry of the ACIST Cardiovascular Pressure Measurement (CPM) System and Navvus Catheter in Clinical Practice-ADVANCE-EU
Brief Title: Post-Market Registry of the ACIST CPM System and Navvus Catheter in Clinical Practice
Acronym: ADVANCE-EU
Status: Completed | Type: Observational
Sponsor: Acist Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: EU100
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Rapid Exchange; Catheter
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Navvus Catheter FFR: The Navvus Catheter is a rapid exchange microcatheter with a pressure sensor at the distal tip that measures Fractional Flow Reserve measurements to guide PCI treatment strategy.
  Interventions: Device: Navvus Catheter FFR

INTERVENTIONS:
Device: Navvus Catheter FFR — Navvus Catheter provides Fractional Flow Reserve (FFR) measurement for each lesion identified according to standard of care of the center and the Instructions for Use (IFU).

SUMMARY:
This registry will collect real-world clinical evidence on the performance, safety, and usability of the ACIST CPM System and NAVVUS Catheter when used in accordance with approved labeling in a European commercial setting. Up to 60 subjects will have Fractional Flow Reserve (FFR) measurements of coronary lesions attempted with the CPM System and NAVVUS Catheter. All subjects will receive diagnostic treatment according to clinical indications and center standard practice.

DETAILED DESCRIPTION:
There are no protocol-specific procedural requirements for this registry. Enrolled subjects will undergo a diagnostic angiography procedure including an FFR measurement with the CPM System and NAVVUS Catheter according to the center standard of care and the Instructions for Use of the CPM System and Navvus Catheter. Participants will be followed for the duration of hospital stay, an expected average of 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older in whom FFR measurement is indicated to guide percutaneous coronary intervention (PCI) strategy and use of the ACIST CPM System and Navvus Catheter is attempted.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older, in whom FFR measurement is indicated to guide PCI strategy and use of the ACIST CPM System and Navvus Catheter is attempted.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Procedural Success | From enrollment through hospital discharge, an expected average of 1 day.
  Procedural success is defined as the ability of the ACIST CPM System and NAVVUS Catheter to acquire FFR measurement without adverse device effect or device malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lefèvre, MD, Principal Investigator — Hospital Privé Jacques Cartier
Locations (7):
- France (2):
  - Hospital Privé Jacques Cartier, Massy
  - Centre Cardiologique du Nord, Saint-Denis
- Germany (3):
  - Johann Wolfgang Goethe Universität, Frankfurt
  - Klinikum Fulda gAG, Fulda
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Ospedale San Raffaele, Milan, Italy
- Hospital Universitario San Juan de Alicante, Alicante, Spain